CLINICAL TRIAL: NCT03788356
Title: Acute Effects of Inspiratory Muscle Training at Different Intensities in Healthy People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Buse Ozcan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/14-16
Record Dates: First submitted 2018-12-18; First posted 2018-12-27 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diaphragmatic breathing (Experimental): Diaphragmatic breathing exercise for 15 minutes.
  Interventions: Other: Diaphragmatic breathing
- 10% inspiratory muscle training (Experimental): Inspiratory muscle training at 10% intensity of maximal inspiratory pressure for 15 minutes
  Interventions: Device: Inspiratory muscle training
- 30% inspiratory muscle training (Experimental): Inspiratory muscle training at 30% intensity of maximal inspiratory pressure for 15 minutes
  Interventions: Device: Inspiratory muscle training
- 60% inspiratory muscle training (Experimental): Inspiratory muscle training at 60% intensity of maximal inspiratory pressure for 15 minutes
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Inspiratory muscle training with a device
  Arms: 10% inspiratory muscle training; 30% inspiratory muscle training; 60% inspiratory muscle training
Other: Diaphragmatic breathing — Diaphragmatic breathing exercise
  Other Names: Exercise
  Arms: Diaphragmatic breathing

SUMMARY:
At least 30 volunteers will be included in the study. After questioning the demographic and clinical information of the participants, dyspnea perception, respiratory functions, respiratory muscle strength, heart rate variability, arterial stiffness, and blood pressure and physical activity levels will be evaluated. Inspiratory muscle training will be done for 15 minutes with an electronic device. Respiratory training will be applied at three different concentrations with 10%, 30% and 60% of maximal inspiratory pressure. Heart rate variability, arterial stiffness, and blood pressure measurements will be repeated after inspiratory muscle training sessions at different intensities.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of mortality in developed and developing countries and constitute a significant morbidity burden for life. Cardiovascular diseases risk factors include obesity, lipid profile, unhealthy diet, sedentary lifestyle, high blood pressure, increased arteriosclerosis.

Although aerobic exercise is recommended as exercise modality to reduce cardiovascular risk, the effects of resistant exercise on cardiovascular health are not clear. In addition, regular aerobic and resistant exercise regulate cardiac autonomic function.

Inspiratory muscle training is a time-efficient, well-tolerated and safe approach for both healthy people and people with chronic diseases. Long-term inspiratory muscle training has been shown to increase respiratory muscle strength and decrease blood pressure in healthy individuals. One-session inspiratory muscle training has been shown to improve autonomic function in smokers and older individuals. However, the effects of different intensities of inspiratory muscle training on blood pressure, autonomic function, and arterial stiffness in healthy young people are not fully understood. For these reasons, the aim of the study is to investigate the acute effects of inspiratory muscle training at different intensities in healthy people.

At least 30 volunteers will be included in the study. After questioning the demographic and clinical information of the participants, dyspnea perception, respiratory functions, respiratory muscle strength, heart rate variability, arterial stiffness, and blood pressure and physical activity levels will be evaluated. Inspiratory muscle training will be done for 15 minutes with an electronic device. Respiratory training will be applied at three different concentrations with 10%, 30% and 60% of maximal inspiratory pressure. Heart rate variability, arterial stiffness, and blood pressure measurements will be repeated after inspiratory muscle training sessions at different intensities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy People

Exclusion Criteria:

* Body mass index (BMI) > 30 kg/m²
* Smoking
* The presence of exercise habit
* Medication use
* Neurological, cardiovascular or respiratory disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Change from Baseline at 15 minutes
  The heart rate is the number of beats per minute of the heart. It represents both sympathetic and parasympathetic system activity. increased heart rate indicates that the sympathetic activity is dominant, while decreased heart rate indicates that parasympathetic activity is dominant.
Augmentation Index | Change from Baseline at 15 minutes
  Augmentation index is commonly used noninvasive measurements of wave reflection strength. To assess augmentation index, brachial artery compression waveforms were obtained by partially inflating a cuff over the brachial artery approximately midway between the shoulder and the elbow. The brachial waveforms were calibrated using cuff-measured brachial systolic and diastolic pressures, and then used to generate central aortic pressure waveforms by applying proprietary digital signal processing and transfer function. The central aortic pulse wave was used to determine augmentation index. High values represent abnormal wave reflection strength.
Aortic Pulse Wave Velocity | Change from Baseline at 15 minutes
  Aortic pulse wave velocity is commonly used noninvasive measurements of arterial stiffness. To assess aortic pulse wave velocity, carotid pulse waves were measured by applanation tonometry and femoral pulse waves were simultaneously obtained by a partially inflated cuff over the femoral artery at the leg midway between the hip and the knee. Aortic pulse wave velocity was determined by calculating the ratio of the corrected distance between the pulse measuring sites to the time delay between the carotid and femoral pulse waves. High values represent increased arterial stiffness.
Square Root of The Mean Squared Difference of Successive Normal to Normal R-R Intervals | Change from Baseline at 15 minutes
  Square Root of The Mean Squared Difference of Successive Normal to Normal R-R Intervals is one of the time domain methods of heart rate variability. It represents a primarily parasympathetic activity or vagal modulation. Low values indicate decreased parasympathetic activity. High values indicate increased parasympathetic activity.

SECONDARY OUTCOMES:
Maximal inspiratory pressure | At Baseline
  Assessment of maximal inspiratory pressure with an electronic mouth pressure device (Micro; Micro Medical Ltd., Rochester, UK). Higher values indicate stronger inspiratory muscle strength.
Maximal expiratory pressure | At Baseline
  Assessment of maximal expiratory pressure with an electronic mouth pressure device (Micro; Micro Medical Ltd., Rochester, UK). Higher values indicate stronger expiratory muscle strength.
Blood pressure | Change from Baseline at 15 minutes
  Brachial and central systolic and diastolic blood pressure. High Brachial and central systolic and diastolic blood pressure are associated with higher risk of heart attacks and strokes, even in people with normal cuff Blood pressure.
Forced vital capacity | At Baseline
  Forced vital capacity is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Vital capacity | At Baseline
  The vital capacity is the volume of air a subject is able to expire after a maximal inspiration to the total lung capacity.
Forced expiratory volume in 1 second | At Baseline
  The volume of air expired in the first second of expiration or forced expiratory volume in 1 second, especially when expressed as a ratio with the total amount of air expired during the forced vital capacity, is a good index of expiratory airways resistance.
International Physical Activity Questionnaire | At Baseline
  The International Physical Activity Questionnaire short-form measures physical activity. The International Physical Activity Questionnaire short-form occurs 7 items. The higher values indicate better physical activity level. The minimum score of scale was 0, and maximum score is depend on patients activity and there is no maximum score.
Fatigue level | Change from Baseline at 15 minutes
  Fatigue level after the training will be questioned with a 100-mm visual analog scale, minimum 0 to maximum 100. Higher scores indicate higher fatigue levels.
Dyspnea level | Change from Baseline at 15 minutes
  Dyspnea level after the training will be questioned with the modified Borg Scale. Minimum value is 0 (no dyspnea), and maximum value is 10 (maximal dyspnea) Higher scores indicate higher fatigue levels.
Percentage Of Successive N-N Intervals With A Difference of Duration Longer Than 50 ms | Change from Baseline at 15 minutes
  Square Root of The Mean Squared Difference of Successive Normal to Normal R-R Intervals is one of the time domain methods of heart rate variability. It represents parasympathetic activity. Low values indicate decreased parasympathetic activity. High values indicate increased parasympathetic activity.
Low Frequency Power | Change from Baseline at 15 minutes
  Low Frequency is one of the frequency domain methods of heart rate variability. Spectral power analysis is performed on a series of R-R intervals which separates the heart rate spectrum into various components and allows the quantification of sympathetic and vagal influences on the heart. Low Frequency range is 0.04-0.15 Hz. Low frequency band represents both sympathetic and parasympathetic modulation.
High Frequency Power | Change from Baseline at 15 minutes
  High Frequency is one of the frequency domain methods of heart rate variability. Spectral power analysis is performed on a series of R-R intervals which separates the heart rate spectrum into various components and allows the quantification of sympathetic and vagal influences on the heart. High Frequency range is 0.15-0.4 Hz. High Frequency band represents parasympathetic modulation. Low values indicate decreased parasympathetic activity. High values indicate increased parasympathetic activity.
Low Frequency/High Frequency ratio | Change from Baseline at 15 minutes
  Low Frequency/High Frequency ratio is one of the frequency domain methods of heart rate variability. Low Frequency/High Frequency ratio is a index of sympathovagal balance. Increased ratio indicates that the sympathetic activity is dominant, while decreased ratio indicates that parasympathetic activity is dominant.
Total Power | Change from Baseline at 15 minutes
  Total Power is one of the frequency domain methods of heart rate variability. It shows general change of autonomic modulation. Low values indicate decreased autonomic modulation. High values indicate increased autonomic modulation.
Pulse Transit Time | Change from Baseline at 15 minutes
  Pulse transit time is the time that takes the pulse pressure wave to travel through the arterial tree. Decreased pulse transit time shows increased wave velocity on the vessels.
Standard Deviation of Normal to Normal R-R Intervals | Change from Baseline at 15 minutes
  Standard Deviation of Normal to Normal R-R Intervals is one of the time domain methods of heart rate variability. Time Domain Analysis measures the change in heart rate over time or the intervals between successive normal cardiac cycles.It assesses globally heart rate variability. Low values indicate decreased heart rate variability. High values indicate increased heart rate variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tanriverdi A, Kahraman BO, Ozsoy I, Ozpelit E, Savci S. Acute effects of inspiratory muscle training at different intensities in healthy young people. Ir J Med Sci. 2021 May;190(2):577-585. doi: 10.1007/s11845-020-02353-w. Epub 2020 Aug 26. PMID 32851483